CLINICAL TRIAL: NCT03056820
Title: Comparison of Apnea Tolerance in Two Positions of Patients With Body Mass Index (BMI) 30-40
Brief Title: Comparison of Apnea Tolerance in Two Positions of Patients With BMI 30-40
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12197
Record Dates: First submitted 2017-01-27; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: General Surgery
Keywords: tracheal intubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person measuring and recording the study data will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - 25° head-up position (Active Comparator): Participants will be positioned at 25° angle for procedure.
  Interventions: Other: 25° head-up position
- B - 55° head-up position (Active Comparator): Participants will be positioned at 55° angle for procedure.
  Interventions: Other: 55° head-up position

INTERVENTIONS:
Other: 25° head-up position — Participant will be positioned at 25° angle for procedure.
  Arms: A - 25° head-up position
Other: 55° head-up position — Participant will be positioned at 55° angle for procedure.
  Arms: B - 55° head-up position

SUMMARY:
The purpose of this study is to compare the effect of the 25° head-up position versus the 55° head-up position on tolerable apnea time (TAT) after induction of general anesthesia in patients with a body mass index (BMI) of 30-40.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* Body Mass Index (BMI) of 30-40
* Scheduled for an elective surgery that requires tracheal intubation

Exclusion Criteria:

* Patients with abnormalities of the upper airway that require awake tracheal intubation
* Asthma
* Chronic obstructive pulmonary disease
* Congestive heart failure
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Tolerable Apnea Time (TAT) | Time between start of induction of general anesthesia (SpO2 100%) to decline of SpO2 94%, up to eight minutes
  Measure of the TAT between groups to determine if the TAT is a function of the participant's position.

SECONDARY OUTCOMES:
Length of time to intubation (TTI) | Time between start of the tracheal intubation procedure to completion of tracheal intubation, up to 2 minutes
Peripheral arterial hemoglobin oxygen saturation (SpO2) trough | Time until SpO2 decreased to 92%, up to 8 minutes
  Measure of the rebound SpO2. It is the lowest SpO2 reading reached subsequent to start of mechanical ventilation at the SpO2 value of 94% and it represents final completion of SpO2 decline.

CONTACTS AND LOCATIONS:
Overall Officials: Mirsad Dupanović, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States